CLINICAL TRIAL: NCT05015049
Title: An Investigation of the Neonatal Burden of Disease of Hypertensive Disorders of Pregnancy: a Population-based Study Using the National Neonatal Research Database
Brief Title: Hypertensive Disorders of Pregnancy - the Neonatal Burden of Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 295875
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal population - hypertensive disorder of pregnancy: All babies born to a woman with a hypertensive disorder of pregnancy (HDP) and admitted to a neonatal unit in England and Wales between 1st January 2012 and 31st December 2020
- Neonatal population - no hypertensive disorder of pregnancy: All babies born to a woman without a hypertensive disorder of pregnancy (HDP) and admitted to a neonatal unit in England and Wales between 1st January 2012 and 31st December 2020

SUMMARY:
Around one in ten women have high blood pressure in pregnancy. This is potentially serious, with risks to the woman and her baby. Whilst maternal deaths from high blood pressure in pregnancy are now rare in the UK, blood pressure problems in pregnancy still cause many stillbirths and early births. Studies have shown that women of Black and Asian backgrounds are more likely to have worse pregnancy outcomes when blood pressure problems in pregnancy develop.

This study aims to:

i) describe the burden of disease of high blood pressure in pregnancy amongst babies admitted to neonatal units on a national scale.

ii) investigate outcomes for babies born to women with high blood pressure in pregnancy admitted to UK neonatal units across maternal ethnic groups.

To complete this study, we will use the National Neonatal Research Database, which holds population-level data for all babies admitted to neonatal units (where unwell babies receive care) in the UK. We will look at records of babies admitted to neonatal units in England and Wales between 2012 and 2020. The records will include information on over half a million babies and their mothers. We will assess how many babies admitted to neonatal units were born to women who had high blood pressure in pregnancy. We will report the outcomes of these babies, and how they compare to babies born to women without high blood pressure in pregnancy. We will analyse whether outcomes for babies born to women with high blood pressure in pregnancy varies according to maternal ethnicity, and investigate what may be driving differences we find.

DETAILED DESCRIPTION:
Study Aims

This study aims to:

* quantify the proportion of all babies admitted to neonatal units born to women with a hypertensive disorder of pregnancy
* describe the national neonatal morbidity, mortality and resource use of babies admitted to neonatal units born to women with a hypertensive disorder of pregnancy
* examine ethnic disparities in neonatal outcomes of babies admitted to neonatal units born to women with hypertensive disorders of pregnancy.

The National Neonatal Research Database (NNRD)

The NNRD is an approved research database constituting real-world prospective clinical data extracted from point-of-care neonatal electronic health records with complete coverage of infants admitted for neonatal care to National Health Service (NHS) neonatal units in England and Wales (since 2012) and Scotland (since 2015). A defined data extract of approximately 450 items (the Neonatal Data Set) is transmitted quarterly to the Neonatal Data Analysis Unit at Imperial College London for data linkage and cleaning prior to entry into the NNRD. To date, the NNRD contains data for over a million babies (approximately 80,000 babies annually). High completeness and accuracy (>95%) of neonatal data held in the NNRD has been confirmed by formal comparison with a multicentre, randomised placebo-controlled trial.

Study Design

This study is a secondary analysis of an existing national electronic health record population cohort using anonymised, routinely recorded clinical data from the National Neonatal Research Database (NNRD). There will be no new patients recruited and there will be no changes made to patient care.

The research team will work with NNRD data analysts to extract anonymised data from the NNRD. A cohort of babies born to women with a hypertensive disorder of pregnancy (HDP) will be defined based on records of maternal medical problems prior to pregnancy, obstetrics problems during pregnancy, medications given during labour and neonatal discharge diagnoses. The morbidity, mortality and health resource use of this cohort will be described in depth. This cohort will also be compared to a cohort of babies born to women without a hypertensive disorder of pregnancy. The HDP cohort will also be stratified by maternal ethnicity to investigate disparities in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must be born between 1st January 2012 and 31st December 2020
* Must be admitted to and received all care in a National Health Service (NHS) neonatal unit in England or Wales

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Babies born between 1st January 2012 and 31st December 2020 and admitted to a neonatal unit in England or Wales
Sampling Method: Probability Sample
Enrollment: 823957 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Survival to discharge from neonatal care | From birth to discharge or death, assessed up to 1 year
  Survival to discharge from neonatal care
Primary recorded reason for neonatal unit admission | From birth to discharge or death, assessed up to 1 year
  Primary recorded reason for neonatal unit admission
Length of stay in neonatal unit | From birth to discharge or death, assessed up to 1 year
  Length of stay in neonatal unit
Number of days of intensive care | From birth to discharge or death, assessed up to 1 year
  Number of days of intensive care

SECONDARY OUTCOMES:
Survival to discharge from neonatal care without comorbidity | From birth to discharge or death, assessed up to 1 year
  Survival to discharge from neonatal care without comorbidity
Cause of death | From birth to discharge or death, assessed up to 1 year
  Cause of death
Age at death | From birth to discharge or death, assessed up to 1 year
  Age at death
Discharge weight SDS (standard deviation score) | From birth to discharge or death, assessed up to 1 year
  Discharge weight SDS (standard deviation score)
Birthweight centile (z-score) | From birth to discharge or death, assessed up to 1 year
  Birthweight centile (z-score)
Clinical diagnoses potential specific to hypertensive disorders of pregnancy | From birth to discharge or death, assessed up to 1 year
  Fetal growth restriction/intrauterine growth restriction, hypoglycaemia
General neonatal complications | From birth to discharge or death, assessed up to 1 year
  Brain injury on imaging, necrotising enterocolitis, sepsis, jaundice, GI perforation
Preterm complications | From birth to discharge or death, assessed up to 1 year
  Chronic lung disease/bronchopulmonary dysplasia, retinopathy of prematurity
Number of days of high-dependancy care | From birth to discharge or death, assessed up to 1 year
  Number of days of high-dependancy care
Number of days of special care | From birth to discharge or death, assessed up to 1 year
  Number of days of special care
Number of days of invasive respiratory support | From birth to discharge or death, assessed up to 1 year
  Number of days of invasive respiratory support
Number of days of non-invasive respiratory support | From birth to discharge or death, assessed up to 1 year
  Number of days of non-invasive respiratory support
Transfusion of blood products | From birth to discharge or death, assessed up to 1 year
  Transfusion of blood products
Number of days of parenteral nutrition | From birth to discharge or death, assessed up to 1 year
  Number of days of parenteral nutrition
Method of feeding (number of days of each e.g. NG, breast etc) | From birth to discharge or death, assessed up to 1 year
  Method of feeding (number of days of each e.g. NG, breast etc)
Type of feeding (number of days of each e.g. breastmilk, formula etc) | From birth to discharge or death, assessed up to 1 year
  Type of feeding (number of days of each e.g. breastmilk, formula etc)
Number of days nil by mouth | From birth to discharge or death, assessed up to 1 year
  Number of days nil by mouth
Line type(s) | From birth to discharge or death, assessed up to 1 year
  Line type(s)
Surfactant administered | From birth to discharge or death, assessed up to 1 year
  Surfactant administered
Surfactant administered on first day | From birth to discharge or death, assessed up to 1 year
  Surfactant administered on first day

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Battersby, Principal Investigator — Imperial College London; Lucy Chappell, Principal Investigator — King's College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided